CLINICAL TRIAL: NCT05093426
Title: Personalised Electronic Record Supported Two-Stage Observational Study of Sleep in Patients With Breast Cancer
Brief Title: PERSONAL - Sleep In Breast Cancer
Status: Completed | Type: Observational
Sponsor: Closed Loop Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: CLM-INS-004
Record Dates: First submitted 2021-09-29; First posted 2021-10-26 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Insomnia; Breast Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Insomnia in Breast cancer cohort: A single cohort will be observed in Stage 1 to assess the prevalence of insomnia suffered by participants who suffer from breast cancer. A subset of participants will continue to Stage 2 to use a digital sleep diary app for an observational period of 3 weeks.
  Interventions: Other: Stage 2 Digital sleep diary app

INTERVENTIONS:
Other: Stage 2 Digital sleep diary app — Participants in Stage 2 will be asked to download a digital sleep diary app and complete a sleep log every day for 21 days.

SUMMARY:
Sleep is essential for human function, immunity, and well-being. In the general population, sleep disturbance and insomnia cause significant health problems and impact on the quality of life of many individuals. The incidence of insomnia in cancer patients is disproportionality higher, with breast cancer patients experiencing prevalence rates ranging from 19% to 69%. The impact of insomnia on cancer patients' lives can be significant and is associated with depression, cancer-related fatigue, increased pain, reduced quality of life, decreased immunity, disease progression, and survival. To date, breast cancer studies show large variation in reported insomnia prevalence rates, and the severity of sleep complaints in these patients have been difficult to assess. Thus, these issues require further investigation using standardised and validated measures.

In this observational study, we aim to investigate the prevalence and severity of insomnia in a cohort of breast cancer patients at the Christie Hospital using the Insomnia Severity Index (ISI), a validated measure for insomnia. This study will consist of two stages. In Stage 1, patients aged 18 and over, who provide informed consent and have a diagnosis of Stage I, II or III breast cancer in the previous 12 months will be asked to complete the validated ISI. Using the ISI, participants identified as having sleeping difficulties and/or insomnia will be invited to Stage 2 of the study. In this stage, participants will be asked to track their sleep each morning for 3 weeks using a digital sleep diary downloaded onto their own smartphone. They will also be asked to complete a series of questionnaires gathering information regarding their quality of life, well-being, and health. This research will provide a better understanding of sleeping patterns, sleeping difficulties and insomnia in patients with breast cancer, and in the long-term, help us design better treatments for patients with sleeping problems.

ELIGIBILITY:
Inclusion Criteria

Stage 1:

* Age > 18 years.
* Informed consent to Stage 1 of the study
* Diagnosis of Stage I, II or III breast cancer within the previous 12 months

Stage 2:

* Informed consent to Stage 2 of the study
* Current Sleep Disturbance; a score of 8 or more on the Insomnia Severity Index.
* History of sleep disturbance prior to the screening/baseline consultation; with beginning or worsening of sleep disturbance since breast cancer diagnosis e.g. sleep problems began or get worse with the diagnosis of breast cancer or with chemotherapy.
* Possession of a suitable smartphone that participant can use independently.

Exclusion Criteria:

Stage 1:

* Participants who have limited or no understanding of spoken and/or written English.
* Other diagnosis of cancer, not including basal cell carcinoma of the skin or cervical carcinoma in situ, within the previous 5 years

Stage 2:

* Co-morbidities incompatible with study participation e.g. that result in a participant being unable to complete daily entries satisfactorily via his/her smartphone.
* Known and/or treated sleep apnoea
* Regular shift work or night work (defined as >1 overnight shift per month)
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of patients diagnosed with breast cancer in the United Kingdom.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Armstrong, PhD, MRCP, MBChB, BSc(Hons), Principal Investigator — Christie NHS Foundation Trust
Locations (1):
- Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed whether the individual participant data will be shared

REFERENCES:
- [Background] Ruel S, Ivers H, Savard MH, Gouin JP, Lemieux J, Provencher L, Caplette-Gingras A, Bastien C, Morin CM, Couture F, Savard J. Insomnia, immunity, and infections in cancer patients: Results from a longitudinal study. Health Psychol. 2020 May;39(5):358-369. doi: 10.1037/hea0000811. Epub 2019 Dec 19. PMID 31855038
- [Background] Kwak A, Jacobs J, Haggett D, Jimenez R, Peppercorn J. Evaluation and management of insomnia in women with breast cancer. Breast Cancer Res Treat. 2020 Jun;181(2):269-277. doi: 10.1007/s10549-020-05635-0. Epub 2020 Apr 20. PMID 32314110
- [Background] Fleming L, Randell K, Stewart E, Espie CA, Morrison DS, Lawless C, Paul J. Insomnia in breast cancer: a prospective observational study. Sleep. 2019 Mar 1;42(3):zsy245. doi: 10.1093/sleep/zsy245. PMID 30521041
- [Background] Fontes F, Pereira S, Costa AR, Goncalves M, Lunet N. The impact of breast cancer treatments on sleep quality 1 year after cancer diagnosis. Support Care Cancer. 2017 Nov;25(11):3529-3536. doi: 10.1007/s00520-017-3777-6. Epub 2017 Jun 16. PMID 28623402
- [Background] Fortner BV, Stepanski EJ, Wang SC, Kasprowicz S, Durrence HH. Sleep and quality of life in breast cancer patients. J Pain Symptom Manage. 2002 Nov;24(5):471-80. doi: 10.1016/s0885-3924(02)00500-6. PMID 12547047
- [Background] Hajj A, Hachem R, Khoury R, Nehme T, Hallit S, Nasr F, Karak FE, Chahine G, Kattan J, Khabbaz LR. Clinical and Genetic Factors Associated With the Breast Cancer-Related Sleep Disorders: The "CAGE-Sleep" Study-A Cross-Sectional Study. J Pain Symptom Manage. 2021 Sep;62(3):e46-e55. doi: 10.1016/j.jpainsymman.2021.02.022. Epub 2021 Feb 22. PMID 33631331
- [Background] Savard J, Ivers H, Villa J, Caplette-Gingras A, Morin CM. Natural course of insomnia comorbid with cancer: an 18-month longitudinal study. J Clin Oncol. 2011 Sep 10;29(26):3580-6. doi: 10.1200/JCO.2010.33.2247. Epub 2011 Aug 8. PMID 21825267
- [Background] Brzecka A, Sarul K, Dyla T, Avila-Rodriguez M, Cabezas-Perez R, Chubarev VN, Minyaeva NN, Klochkov SG, Neganova ME, Mikhaleva LM, Somasundaram SG, Kirkland CE, Tarasov VV, Aliev G. The Association of Sleep Disorders, Obesity and Sleep-Related Hypoxia with Cancer. Curr Genomics. 2020 Sep;21(6):444-453. doi: 10.2174/1389202921999200403151720. PMID 33093806
- [Background] Palesh O, Aldridge-Gerry A, Zeitzer JM, Koopman C, Neri E, Giese-Davis J, Jo B, Kraemer H, Nouriani B, Spiegel D. Actigraphy-measured sleep disruption as a predictor of survival among women with advanced breast cancer. Sleep. 2014 May 1;37(5):837-42. doi: 10.5665/sleep.3642. PMID 24790261
- [Background] Savard J, Morin CM. Insomnia in the context of cancer: a review of a neglected problem. J Clin Oncol. 2001 Feb 1;19(3):895-908. doi: 10.1200/JCO.2001.19.3.895. PMID 11157043
- [Background] Marion LP, Ivers H, Savard J. Feasibility of a Preventive Intervention for Insomnia in Women with Breast Cancer Receiving Chemotherapy. Behav Sleep Med. 2021 Jan-Feb;19(1):70-82. doi: 10.1080/15402002.2019.1707203. Epub 2019 Dec 24. PMID 31873040
- [Background] O'Donnell JF. Insomnia in cancer patients. Clin Cornerstone. 2004;6 Suppl 1D:S6-14. doi: 10.1016/s1098-3597(05)80002-x. PMID 15675652
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Horsch CH, Lancee J, Griffioen-Both F, Spruit S, Fitrianie S, Neerincx MA, Beun RJ, Brinkman WP. Mobile Phone-Delivered Cognitive Behavioral Therapy for Insomnia: A Randomized Waitlist Controlled Trial. J Med Internet Res. 2017 Apr 11;19(4):e70. doi: 10.2196/jmir.6524. PMID 28400355
- [Background] Kang SG, Kang JM, Cho SJ, Ko KP, Lee YJ, Lee HJ, Kim L, Winkelman JW. Cognitive Behavioral Therapy Using a Mobile Application Synchronizable With Wearable Devices for Insomnia Treatment: A Pilot Study. J Clin Sleep Med. 2017 Apr 15;13(4):633-640. doi: 10.5664/jcsm.6564. PMID 28162145
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Fallowfield LJ, Leaity SK, Howell A, Benson S, Cella D. Assessment of quality of life in women undergoing hormonal therapy for breast cancer: validation of an endocrine symptom subscale for the FACT-B. Breast Cancer Res Treat. 1999 May;55(2):189-99. doi: 10.1023/a:1006263818115. PMID 10481946
- See also: Epidemiology of Insomnia - Prevalence, Course, Risk Factors, and Public Health Burden — https://doi.org/10.1016/j.jsmc.2013.05.002
- See also: Insomnia in breast cancer: prevalence and associated factors — http://dx.doi.org/10.1136/bmjspcare-2020-002718
- See also: Disruption of sleep, sleep-wake activity rhythm, and nocturnal melatonin production in breast cancer patients undergoing adjuvant chemotherapy: a prospective cohort study — https://doi.org/10.1016/j.sleep.2018.11.022
- See also: Joint statement on seeking consent by electronic methods — https://s3.eu-west-2.amazonaws.com/www.hra.nhs.uk/media/documents/hra-mhra-econsent-statement-sept-18.pdf
- See also: Consent and Participant Information Guidance — http://www.hra-decisiontools.org.uk/consent/
- See also: Sample Size Calculator for Estimating a Single Proportion — https://statulator.com/SampleSize/ss1P.html
- See also: Construction and Evaluation of a User Experience Questionnaire — https://doi.org/10.1007/978-3-540-89350-9_6

RESULTS

PARTICIPANT FLOW:
Period: Stage 1
Arm/Group | Insomnia in Breast Cancer Cohort
Started | 226
Completed | 220
Not Completed | 6
Period: Stage 2
Arm/Group | Insomnia in Breast Cancer Cohort
Started | 120
Completed | 105
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 missing values
  years
    number analyzed (Participants) | 218
    (all) | 53.9 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Female | 218
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    Ethnicity: number analyzed (Participants) | 218
    Ethnicity: Asian/British Asian | 6
    Ethnicity: Black/African/Black British | 5
    Ethnicity: Mixed/Multiple ethnic backgrounds | 4
    Ethnicity: Other ethnic group | 1
    Ethnicity: White | 202
Smartphone access [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Yes | 214
    No | 4
Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: 2 missing values
  kg
    number analyzed (Participants) | 218
    (all) | 76.1 (16.68)
Height (cm) [Mean (Standard Deviation); unit: cm] — Population: 2 missing values
  cm
    number analyzed (Participants) | 218
    (all) | 163.5 (7.33)
Body Mass Index (kg/m^2) [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Underweight | 3
    Normal weight | 68
    Overweight | 74
    Obese | 59
    Morbidly obese | 14
Breastfeeding [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    (all) | 218
Regular night-work/shift work [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Yes | 2
    No | 216
Marital status [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Married or living with partner | 163
    Separated or divorced | 27
    Single | 22
    Widowed | 6
Education level [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    College | 67
    Primary school | 1
    Secondary school | 48
    University | 102
Employment status [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Full-time work | 111
    Part-time work | 52
    Retired | 42
    Student | 1
    Unemployed | 12
Menopausal status [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Don't know | 26
    Peri-menopause | 37
    Post-menopause | 123
    Pre-menopause | 32
Sleep difficulties [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Yes | 168
    No | 50
Sleep difficulties started/worsened since diagnosis [Count of Participants; unit: Participants] — Population: 16 missing values
  Participants
    number analyzed (Participants) | 204
    Yes | 150
    No | 54
Prescribed medication for sleep issues [Count of Participants; unit: Participants] — Population: 52 missing values
  Participants
    number analyzed (Participants) | 168
    Yes | 12
    No | 156
Sleep apnoea [Count of Participants; unit: Participants] — Population: 2 missing values
  Participants
    number analyzed (Participants) | 218
    Yes | 3
    No | 215

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Insomnia in a Cohort of Breast Cancer Patients
Description: Percentage of breast cancer patients scoring 8 or above on the Insomnia Severity Index
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 220
Participants | 170

2. Secondary Outcome: In Patients With Breast Cancer Experiencing Insomnia (Defined as Score of 8 or More on the Insomnia Severity Index; ISI Scale), to Assess Insomnia Severity Over a Three-week Period.
Description: Insomnia severity using Insomnia Severity Index (min. 0, max. 28 where higher scores mean a worse outcome). With severity classified by total score for the Insomnia Severity Index: 0-7 no significant insomnia, 8-14 Subthreshold insomnia, 15-21 Clinical insomnia (moderate severity) and 22-28 Clinical Insomnia (Severe severity)
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 220
Participants
  No clinically significant insomnia | 50
  Subthreshold insomnia | 90
  Clinical insomnia (moderate severity) | 71
  Clinical insomnia (severe) | 9

3. Secondary Outcome: In Patients With Breast Cancer Experiencing Insomnia (Defined as Score of 8 or More on the Insomnia Severity Index; ISI Scale), to Assess Sleep Efficiency Over a Three-week Period.
Description: In patients with breast cancer experiencing insomnia (defined as score of 8 or more on the Insomnia Severity Index; ISI scale), to assess Sleep efficiency over a three-week period. Sleep efficiency (the % of time a participant is asleep whilst in bed) measured using Sleep diary (derived from total time asleep relative to total time in bed).
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: percentage of time participant is asleep
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 97
percentage of time participant is asleep | 78.5 (10.71)

4. Secondary Outcome: In Patients With Breast Cancer Experiencing Insomnia (Defined as Score of 8 or More on the Insomnia Severity Index; ISI Scale), to Assess Quality of Life Over a Three-week Period.
Description: Quality of Life using EQ-5D-5L questionnaire (multiple choice questions regarding Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression as well as measure of % of health using scale where higher percentage is greater outcome) and Functional Assessment of Cancer Therapy - Endocrine Systems questionnaire (questions regarding Physical well-being, Social/Family well-being, Emotional, Functional well-being and Additional concerns using scale of 0 - 4 where 0 is Not at all, 1 is A little bit, 2 is Some-what, 3 is Quite a bit and 4 is Very much).
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 105
Participants
  EQ-5D-5L - Mobility - Baseline: No problems | 87
  EQ-5D-5L - Mobility - Baseline: Some problems | 18
  EQ-5D-5L - Mobility - Baseline: Missing | 0
  EQ-5D-5L - Mobility - Day 21: No problems | 60
  EQ-5D-5L - Mobility - Day 21: Some problems | 38
  EQ-5D-5L - Mobility - Day 21: Missing | 7
  EQ-5D-5L - Self-care - Baseline: No problems | 95
  EQ-5D-5L - Self-care - Baseline: Some problems | 10
  EQ-5D-5L - Self-care - Baseline: Missing | 0
  EQ-5D-5L - Self-care - Day 21: No problems | 86
  EQ-5D-5L - Self-care - Day 21: Some problems | 12
  EQ-5D-5L - Self-care - Day 21: Missing | 7
  EQ-5D-5L - Usual activities - Baseline: No problems | 51
  EQ-5D-5L - Usual activities - Baseline: Some problems | 54
  EQ-5D-5L - Usual activities - Baseline: Missing | 0
  EQ-5D-5L - Usual activities - Day 21: No problems | 24
  EQ-5D-5L - Usual activities - Day 21: Some problems | 74
  EQ-5D-5L - Usual activities - Day 21: Missing | 7
  EQ-5D-5L - Pain/discomfort - Baseline: No problems | 31
  EQ-5D-5L - Pain/discomfort - Baseline: Some problems | 74
  EQ-5D-5L - Pain/discomfort - Baseline: Missing | 0
  EQ-5D-5L - Pain/discomfort - Day 21: No problems | 15
  EQ-5D-5L - Pain/discomfort - Day 21: Some problems | 83
  EQ-5D-5L - Pain/discomfort - Day 21: Missing | 7
  EQ-5D-5L - Anxiety/depression - Baseline: No problems | 35
  EQ-5D-5L - Anxiety/depression - Baseline: Some problems | 70
  EQ-5D-5L - Anxiety/depression - Baseline: Missing | 0
  EQ-5D-5L - Anxiety/depression - Day 21: No problems | 30
  EQ-5D-5L - Anxiety/depression - Day 21: Some problems | 68
  EQ-5D-5L - Anxiety/depression - Day 21: Missing | 7

5. Secondary Outcome: In Patients With Breast Cancer Experiencing Insomnia (Defined as Score of 8 or More on the Insomnia Severity Index; ISI Scale), to Assess Quality of Life Over a Three-week Period.
Description: EQ-5D-5L questionnaire: multiple choice questions for Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression and % of health where a higher % is a greater outcome). Functional Assessment of Cancer Therapy - Endocrine Systems (FACT-ES) (sub-scales: Physical well-being, Social/Family well-being, Emotional, Functional well-being and Endocrine symptoms): each question in sub-scales are scored using a scale of 0-4 where 0 is Not at all, 1 is A little bit, 2 is Some-what, 3 is Quite a bit and 4 is Very much. Scores for questions are added to give total baseline and total day 21 score for each sub-scale. Minimum total score is 0 for all sub-scales, the maximum scores are 28 for Physical, Social/Family and Functional well-being sub-scales, 24 for the Emotional well-being sub-scale, 76 for Endocrine symptoms. A lower total score represents better outcomes. FACT-ES = Total of subscale scores (0-184). FACT-G = Total of subscale scores excluding endocrine system (0-108).
Time Frame: 3 weeks
Population: 7 missing values at Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 105
score on a scale
  FACT-ES - Physical well-being - Total Baseline score | 18.9 (5.00)
  FACT-ES - Physical well-being - Total Day 21 Score: number analyzed (Participants) | 98
  FACT-ES - Physical well-being - Total Day 21 Score | 18.5 (5.40)
  FACT-ES - Social/family well-being - Total Baseline score | 17.9 (4.12)
  FACT-ES - Social/family well-being - Total Day 21 score: number analyzed (Participants) | 98
  FACT-ES - Social/family well-being - Total Day 21 score | 17.1 (4.49)
  FACT-ES - Emotional well-being - Total Baseline score | 16.5 (3.78)
  FACT-ES - Emotional well-being - Total Day 21 score: number analyzed (Participants) | 98
  FACT-ES - Emotional well-being - Total Day 21 score | 16.5 (3.86)
  FACT-ES - Functional well-being - Total Baseline score | 13.0 (4.99)
  FACT-ES - Functional well-being - Total Day 21 score: number analyzed (Participants) | 98
  FACT-ES - Functional well-being - Total Day 21 score | 12.9 (5.04)
  FACT-ES - Endocrine Symptom Subscale - Total Baseline score | 54.0 (9.88)
  FACT-ES - Endocrine Symptom Subscale - Total Day 21 score: number analyzed (Participants) | 98
  FACT-ES - Endocrine Symptom Subscale - Total Day 21 score | 53.1 (9.96)
  FACT-ES - Total Baseline score | 120.1 (18.91)
  FACT-ES - Total Day 21 score: number analyzed (Participants) | 98
  FACT-ES - Total Day 21 score | 118.1 (20.85)
  FACT-G - Total Baseline score | 66.2 (12.55)
  FACT-G - Total Day 21 score: number analyzed (Participants) | 98
  FACT-G - Total Day 21 score | 65.0 (14.18)

6. Secondary Outcome: To Assess: - Compliance of Data Entry Into the Digital Sleep Diary - Feasibility and Experience of Patients to Input Data Relating to Their Sleep Into a Mobile Phone Application Daily
Description: Compliance; % of patients completing sleep diary (17 or more days out of 21) Feasibility and User experience; User experience questionnaire.
Time Frame: 3 weeks
Population: Number of subjects completing the digital sleep diary on at least 17 out of 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 105
Participants | 66

7. Secondary Outcome: Associations Between Insomnia Prevalence and Severity as Measured by the Insomnia Severity Index and Quality of Life (EQ-5D-5L and FACT-ES) With Clinical or Treatment Characteristics of Breast Cancer Patients.
Description: Assessment to determine if there is any association or correlation between insomnia prevalence and severity as well as quality of life (using insomnia severity index and EQ-5D-5L and Functional Assessment of Cancer Therapy - Endocrine Systems questionnaires) for patients in subgroups based on clinical or treatment characteristics i.e. breast cancer stage (Stage I, II or III), tumour staging (T1, T2, T3 or DCIS) treatment regimen (Systemic treatment, Dexamethasone treatment, Radiation therapy, Hormonal or Targeted Therapy as well as time since start of chemotherapy and current systemic anti-cancer therapy).
Time Frame: 3 weeks
Population: These are descriptions of the subgroups that were analysed based on breast cancer stage, tumour staging and treatment regimen therefore the reported numbers reflect the number of participants in each subgroup.
Measure: Count of Participants; unit: Participants
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 105
Participants
  Stage I breast cancer participants who reported as having insomnia (ISI score 8 or above) | 26
  Stage II breast cancer participants who reported as having insomnia (ISI score 8 or above) | 58
  Stage III breast cancer participants who reported as having insomnia (ISI score 8 or above) | 21
  Stage I breast cancer participants who reported as having subthreshold insomnia: number analyzed (Participants) | 26
  Stage I breast cancer participants who reported as having subthreshold insomnia | 12
  Stage I breast cancer participants who reported as having clinical insomnia (moderate severity): number analyzed (Participants) | 26
  Stage I breast cancer participants who reported as having clinical insomnia (moderate severity) | 13
  Stage I breast cancer participants who reported as having clinical insomnia (severe): number analyzed (Participants) | 26
  Stage I breast cancer participants who reported as having clinical insomnia (severe) | 1
  Stage II breast cancer participants who reported as having subthreshold insomnia: number analyzed (Participants) | 58
  Stage II breast cancer participants who reported as having subthreshold insomnia | 30
  Stage II breast cancer participants who reported as having clinical insomnia (moderate severity): number analyzed (Participants) | 58
  Stage II breast cancer participants who reported as having clinical insomnia (moderate severity) | 25
  Stage II breast cancer participants who reported as having clinical insomnia (severe): number analyzed (Participants) | 58
  Stage II breast cancer participants who reported as having clinical insomnia (severe) | 3
  Stage III breast cancer participants who reported as having subthreshold insomnia: number analyzed (Participants) | 21
  Stage III breast cancer participants who reported as having subthreshold insomnia | 9
  Stage III breast cancer participants who reported as having clinical insomnia (moderate severity): number analyzed (Participants) | 21
  Stage III breast cancer participants who reported as having clinical insomnia (moderate severity) | 12
  Stage III breast cancer participants who reported as having clinical insomnia (severe): number analyzed (Participants) | 21
  Stage III breast cancer participants who reported as having clinical insomnia (severe) | 0
  Tumour staging T1 participants who reported as having insomnia (ISI score 8 or above) | 43
  Tumour staging T2 participants who reported as having insomnia (ISI score 8 or above) | 47
  Tumour staging T3 participants who reported as having insomnia (ISI score 8 or above) | 14
  Tumour staging DCIS participants who reported as having insomnia (ISI score 8 or above) | 1
  Systemic anti-cancer therapy participants who reported as having insomnia (ISI score 8 or above) | 54
  Dexamethasone treatment participants who reported as having insomnia (ISI score 8 or above) | 12
  Radiation therapy participants who reported as having insomnia (ISI score 8 or above) | 34
  Targeted therapy participants who reported as having insomnia (ISI score 8 or above) | 16
  Hormonal treatment participants who reported as having insomnia (ISI score 8 or above) | 39

8. Secondary Outcome: Safety of the Digital Sleep Diary
Description: Adverse Events and Serious Adverse Events will be collected and summarised.
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Insomnia in Breast Cancer Cohort
Number analyzed (Participants) | 105
participants
  Number of subjects that experienced any Adverse Event | 51
  Related to the Sleep Diary | 0

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Nurses called participants at the end of the 3-week period to ask if they had experienced any adverse events during the 3-week period.
Arm/Group | Insomnia in Breast Cancer Cohort
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 51/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insomnia in Breast Cancer Cohort (N=105)
Fatigue (General disorders) | 20 (20)
Insomnia (Psychiatric disorders) | 14 (14)
Itchy skin on arms (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Edema limbs (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Stinging on left axilla scar (Nervous system disorders) | 1 (1)
Covid-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 9 (9)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Mood changes (Psychiatric disorders) | 1 (1)
Sleep struggles (Psychiatric disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Low mood (Psychiatric disorders) | 1 (1)
Neuropathy in the tips fingers and soles (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Sore skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Dizzy spells (Nervous system disorders) | 1 (1)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Migraines (Nervous system disorders) | 1 (1)
Blisters (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Discomfort on palpation (Skin and subcutaneous tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Pain around radiotherapy site (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Edema - hands and feet (General disorders) | 1 (1)
Joint ache (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain (General disorders) | 2 (2)
Radiating arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent pain (General disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 3 (3)
Cold sore (Infections and infestations) | 1 (1)
Aching legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Aching joints (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT05093426/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT05093426/SAP_001.pdf